CLINICAL TRIAL: NCT03337347
Title: Clinical Significance of Detecting CEA and CK20 mRNA-positive Cells in Colorectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTC_CRC_2017
Record Dates: First submitted 2017-10-26; First posted 2017-11-09 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Cancer; Circulating Tumor Cell
Keywords: Prognostic significance
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CTC/DTC count — The presence of CTCs/DTCs in the peripheral blood and/or bone marrow may identify colorectal cancer patients with high risk of disease recurrence who may benefit from adjuvant therapy.

SUMMARY:
To determine whether the presence of circulating/disseminated tumor cells (CTCs/DTCs) in the blood and bone marrow of colorectal cancer (CRC) patients with localized disease is a negative prognostic factor, and to find correlations with other clinical/pathological disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

- colorectal adenocarcinoma

Exclusion Criteria:

* prior neoadjuvant chemoradiotherapy
* prior colorectal cancer
* cancer duplicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2007-02-28 (Actual); Study Completion 2015-10-23 (Actual)

PRIMARY OUTCOMES:
CEA mRNA positive circulating tumor cells in colorectal cancer patients | 1 day
  The absolute gene expression of carcinoembryonic antigen (CEA mRNA) in circulating tumor cells (CTCs) purified from peripheral blood of patients before colorectal surgery will be measured using real-time RT-PCR method. The CEA gene expression will be normalized per microgram of total mRNA. The cut-off values identifying presence or absence of CEA mRNA positive CTCs in patients was established using the maxstat() function from the maxstat R package as a mode value of estimates obtained for 10 000 random samples. CEA mRNA levels above 190 CEA mRNA copies per microgram of RNA will indicate the presence of the CTCs in the peripheral blood sample.

SECONDARY OUTCOMES:
Cancer specific survival in CTC positive CRC patients | 10 years
  The cancer specific survival in months will be measured from the time of diagnosis to the time of cancer related death. Two groups of patients will be compared:
  A: Patients with the presence of CEA mRNA positive CTCs in peripheral blood before colorectal cancer surgery as described in primary outcome measure.
  B: Patients with the absence of CEA mRNA positive CTCs in peripheral blood before colorectal cancer surgery as described in primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Miloslav Duda, MD, Principal Investigator — University Hospital Olomouc
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Yes
De-identified primary data will be available